CLINICAL TRIAL: NCT05949411
Title: Development of Non-invasive Methods to Study Gut Microbiome - Nutrition - Host Interactions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MICROBOOST
Record Dates: First submitted 2023-04-17; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Screening (Other): D-42 to D-7
  Interventions: Other: Screening visit
- Lactulose (Other): D0
  Interventions: Other: Lactulose test
- Meal 1 (Other): D14+/-7
  Interventions: Other: Administration of standardized meals with characterized dietary fiber content
- Meal 2 (Other): D16+/-7
  Interventions: Other: Administration of standardized meals with characterized dietary fiber content
- Meal 3 (Other): D18+/-7
  Interventions: Other: Administration of standardized meals with characterized dietary fiber content

INTERVENTIONS:
Other: Screening visit — Subjects will be invited to perform the screening visit to sign the informed consent and then to ensure that they are able to participate in this study.
  Arms: Screening
Other: Lactulose test — Fasted subjects (at least 10 hours) will receive on oral load of 10 g of lactulose. Then, exhaled H2 will be measured every 30 minutes during 4 hours.
  Arms: Lactulose
Other: Administration of standardized meals with characterized dietary fiber content — Subjects will receive standardized breakfasts and lunches characterized in terms of dietary fiber content. Urine, saliva, feces samples will be collected. Breath test and gastrointestinal symptoms will be followed during maximum 8h. Subjects will also complete SF36 questionnaire, food diary and stool/transit questionnaire.
  Arms: Meal 1; Meal 2; Meal 3

SUMMARY:
The aim of this study is to develop and validate an adequate protocol of volatolome (volatile metabolites) measurement in breath of human volunteers (18-65 years) to study gut microbiome - nutrition - host interactions in a general healthy population. For this purpose, breath volatile metabolites (BVM) will be analyzed throughout test days in fasting state and after standardized meals using selected ion flow tube mass spectrometry (SIFT-MS). In addition, gut microbial functions linked notably to hydrogen/methane production, carbohydrates utilization (CAZymes), and in the production of other volatile metabolites of interest (i.e. indole, fatty acid derivatives, ...) will be unraveled through microbiome sequencing data analysis (in silico), metabolomic analyses and measurement of enzymatic activities from saliva, urine and/or fecal samples.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man, aged of 18 to 65 years;
* Body mass index (BMI) between 18 and 30 kg/m2;
* Non-smoker;
* Provision of signed and dated informed consent form;
* Stated willingness to comply with all study procedures and availability for the duration of the study;
* Speaking French.

Exclusion Criteria:

* Subject with severe systemic disease (renal or hepatic failure, cancer, pancreatic cancer, chronic pancreatitis, asthma …)
* Subject with a history or current chronic/severe gastrointestinal disorder such as duodenal ulcer, chronic colitis, or chronic inflammatory disease of the digestive tract disease (Crohn's disease, ulcerative colitis), celiac disease or irritable bowel syndrome;
* Subjects with a history of digestive tract surgery (except appendectomy);
* Subject who had surgery within the two months prior to the study
* Subjects with psychiatric problems and/or using antipsychotics
* Current or recent (< 4 weeks) intake of antibiotics, fiber supplement, and/or any products modulating gut transit (laxative, anti-diarrheal, ...) or gut microbiota composition; these products will also be avoided for the duration of the study;
* Chronic intake of drugs, except contraceptive drug;
* Subject following a low-calorie diet and followed by a doctor or dietician in progress or recently (< 6 weeks);
* Women of childbearing age who are pregnant or breastfeeding or who wish to become pregnant within the next 6 weeks or who are not using an adequate method of contraception (e.g. oral contraception, intrauterine device (IUD), abstinence, ...);
* Subjects who drink more than 3 glasses of alcohol per day (> 30 g of alcohol per day);
* Subjects having participated to another clinical trial two weeks before the screening test visit;
* Subjects who practice an intense sport activity (more than 10 hours per week of intense activity);
* Language barrier, mental or legal incapacity, unwillingness or inability to understand or not being able to participate to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Exhaled volatile compounds | Throughout the entire study, approximately during 24 months
  Selected Ion flow tube mass spectrometry (SIFT-MS) - Area under the curve (calculated on 8 hours following breakfast ingestion)

SECONDARY OUTCOMES:
Gut microbiota | Throughout the entire study, approximately during 24 months
  Illumina sequencing of 16S ribosomal deoxyribonucleic acid (rDNA), quantitative polymerase chain reaction (PCR)
Salivary microbiota | Throughout the entire study, approximately during 24 months
  Illumina sequencing of 16SrDNA, quantitative PCR
Gastrointestinal symptom - discomfort | Throughout the entire study, approximately during 24 months
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 8 hours following breakfast ingestion)
Gastrointestinal symptom - nausea | Throughout the entire study, approximately during 24 months
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 8 hours following breakfast ingestion)
Gastrointestinal symptom - bloating | Throughout the entire study, approximately during 24 months
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 8 hours following breakfast ingestion)
Gastrointestinal symptom - flatulences | Throughout the entire study, approximately during 24 months
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 8 hours following breakfast ingestion)
Gastrointestinal symptom - gastrointestinal reflux | Throughout the entire study, approximately during 24 months
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 8 hours following breakfast ingestion)
Gastrointestinal symptom - cramps | Throughout the entire study, approximately during 24 months
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 8 hours following breakfast ingestion)
Gastrointestinal symptom - rumbling | Throughout the entire study, approximately during 24 months
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 8 hours following breakfast ingestion)
Gastrointestinal symptom - burps | Throughout the entire study, approximately during 24 months
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom)
Gut microbiota metabolic capacity | Throughout the entire study, approximately during 24 months
  Enzymatic analysis via in-vitro studies, incubation of fecal extracts
Exhaled hydrogen (H2) | Throughout the entire study, approximately during 24 months
  Lactotest 202 - Area under the curve (calculated on 4 hours following lactulose ingestion)
Exhaled methane (CH4) | Throughout the entire study, approximately during 24 months
  Lactotest 202 - Area under the curve (calculated on 8 hours following breakfast ingestion)
Exhaled carbon dioxide (CO2) | Throughout the entire study, approximately during 24 months
  Lactotest 202 - Area under the curve (calculated on 4 hours following lactulose ingestion)
Carbohydrates utilization - Carbohydrate active enzymes (CAZymes) | Throughout the entire study, approximately during 24 months
  Saliva enzymatic activities
Nutrient intake | Throughout the entire study, approximately during 24 months
  Food diary (daily log of what the volunteer eats and drinks each day)
Dietary habits | Throughout the entire study, approximately during 24 months
  Food frequency questionnaire (FFQ) (record the volunteers' usual diet and dietary habits)
Well-being | Throughout the entire study, approximately during 24 months
  The short form (36) health survey (SF36) (0 = worse physical and mental health functioning, 100 = best physical and mental health functioning)
Transit - frequency | Throughout the entire study, approximately during 24 months
  Questionnaire on stool frequency (record each defecation time)
Transit - type of stool | Throughout the entire study, approximately during 24 months
  Bristol stools scale (BSS) (classify the form of feces into 7 categories; type 1 = severe constipation, type 2 = mild constipation, types 3 and 4 = normal, type 5 = lacking fiber, type 6 = mild diarrhea, type 7 = severe diarrhea)
Transit - ease of passage | Throughout the entire study, approximately during 24 months
  5-point Likert's scale (1 = very difficult to defecate, 5 = very easy to defecate)
Transit - level of emergency | Throughout the entire study, approximately during 24 months
  5-point Likert's scale (1 = very urgent need to defecate, 5 = very nonurgent need to defecate)
Transit - empty feeling | Throughout the entire study, approximately during 24 months
  5-point Likert's scale (1 = very nonempty feeling after defecation, 5 = very empty feeling after defecation)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Delzenne, Prof., Principal Investigator — Université Catholique de Louvain
Locations (3):
- Belgium (3):
  - Center of Investigation in Clinical Nutrition (CICN), UCLouvain/CICN, Ottignies-Louvain-la-Neuve, Brabant Wallon
  - Metabolism and Nutrition research group (MNUT), Louvain Drug Research Institute (LDRI), UCLouvain, Woluwe-Saint-Lambert, Brussels Capital
  - Testing rooms of Institute of Neuroscience (IONS), UCLouvain/IONS, Woluwe-Saint-Lambert, Brussels Capital

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared by the partners from the Consortium agreement.
  * Gut and salivary microbiota composition;
  * Urinary, salivary and fecal metabolites;
  * Visual analogue scales data;
  * Gut microbial functions;
  * Nutrient intake and dietary habits;
  * Well-being;
  * Transit;
  * Concomitant medication;
  * Inclusion/exclusion criteria;
  * Adverse event.
  Data will be shared at the end of the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the study
Access Criteria: Belonging to the project partner (Consortium agreement)

REFERENCES:
- [Background] Neyrinck AM, Rodriguez J, Zhang Z, Nazare JA, Bindels LB, Cani PD, Maquet V, Laville M, Bischoff SC, Walter J, Delzenne NM. Breath volatile metabolome reveals the impact of dietary fibres on the gut microbiota: Proof of concept in healthy volunteers. EBioMedicine. 2022 Jun;80:104051. doi: 10.1016/j.ebiom.2022.104051. Epub 2022 May 10. PMID 35561452
- [Background] Neyrinck AM, Rodriguez J, Zhang Z, Seethaler B, Mailleux F, Vercammen J, Bindels LB, Cani PD, Nazare JA, Maquet V, Laville M, Bischoff SC, Walter J, Delzenne NM. Noninvasive monitoring of fibre fermentation in healthy volunteers by analyzing breath volatile metabolites: lessons from the FiberTAG intervention study. Gut Microbes. 2021 Jan-Dec;13(1):1-16. doi: 10.1080/19490976.2020.1862028. PMID 33461385